CLINICAL TRIAL: NCT04591678
Title: Characterizing Longitudinal Outcomes in Adults With SMA Treated With Nusinersen
Brief Title: Adults With SMA Treated With Nusinersen
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Biogen (Industry); Cure SMA (Other)
Responsible Party: Principal Investigator, Bakri Elsheikh, Professor of Neurology, Ohio State University
Other Study IDs: 2018H0311
Record Dates: First submitted 2019-10-23; First posted 2020-10-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Spinal Muscular Atrophy
Keywords: nusinersen; Spinraza
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood/serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- SMA nusinersen adult cohort: The nusinersen treatment will be given as standard of care. The treatment (which is NOT research, but the standard care) will be given by an injection into the cerebrospinal fluid (fluid in your spine) through a needle inserted into your lower back. Participants will receive a 12 mg (5 mL) dose during each administration/injection, which will occur on the following days: 1 (baseline), 15, 29, and 60. Following the 60 day treatment, participants will receive treatment every 4 months (6, 10, 14 etc.).
  After the 60 day, 6 month, 10 month, 14 month, 18 month and 22 month treatments the study team will see each participant afterwards to collect information to evaluate your general health, function and response to the treatment for the study.
  Interventions: Drug: nusinersen

INTERVENTIONS:
Drug: nusinersen — SPINRAZA (nusinersen) is FDA approved to treat spinal muscular atrophy (SMA) through intrathecal injection.
  Other Names: SPINRAZA

SUMMARY:
This is a single center, 22-month observational study of nusinersen treatment in adult patients with spinal muscular atrophy (SMA). There will be a total of seven visits. Nusinersen is provided as standard of care and not considered research in this study. Information will be collected regarding the general health, and function including muscle strength of, as well as any positive and/or adverse events experienced by the study participants.

DETAILED DESCRIPTION:
This is a single center, 22-month observational study of nusinersen treatment in adult patients with SMA. There will be a total of five visits. All subjects will be evaluated at a screening visit no more than four weeks before starting their standard of care nusinersen treatment to determine their eligibility for participation. Eligible patients will complete their standard induction intrathecal nusinersen treatment on day 1, 15, 29 and 60 followed by maintenance doses every four months. Subjects will be reevaluated after completing the loading doses at 2 months followed by every four-month evaluations for the total duration of the treatment of 22 months.

Currently, there is no data published on patients receiving this treatment over the age of 18. Without published data collected from research, it is difficult for adult patients to get approval from their insurance companies to receive this treatment. This study hopes to collect data, in order to make this treatment option easier for patients with SMA to access and in general learn how well nusinersen is working in adult patients with SMA overtime.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years
2. Genetic confirmation of 5q SMA documented by the homozygous deletion of both SMN1 genes on standard genetic tests for the disorder
3. SMN2 copy number of 3 or greater
4. Subjects must be able to walk thirty feet without assistance (i.e. no canes, walkers)
5. Interest in participating and the ability to meet the study requirements
6. Women of childbearing-age are required to be on birth control or abstain while participating in the research study

Exclusion Criteria:

1. Subjects with history of spinal disease that will interfere with the lumbar puncture procedure
2. Subjects with history of bacterial meningitis or encephalitis
3. Subjects with history of use of investigational drug treatment for SMA in the last six months, or plan on enrolling in any other treatment trial during the duration of this trial
4. History of treatment with gene therapy, stem cell or antisense oligonucleotide
5. Patients with co-morbid conditions that preclude travel, testing or study medications
6. Patients who are, in the investigator's opinion, mentally or legally incapacitated from providing informed consent for the study, or are otherwise unable to meet study requirements or cooperate reliably with study procedures, especially strength testing
7. Women who are pregnant or who intend to become pregnant while participating in the research study or who are breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with spinal muscular atrophy (SMA) as confirmed by clinical and genetic assessments.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 22 months
  To evaluate the effect of nusinersen treatment on muscle strength in ambulatory SMA adults

SECONDARY OUTCOMES:
Change in Six Minute Walk Test | 22 months
  6 Minute Walk Test (6WMT)
Change in Hammersmith Functional Motor Scale Expanded | 22 months
  Hammersmith Functional Motor Scale Expanded (HFMSE)
Change in SMA Functional Rating Scale | 22 months
  modified SMA Functional Rating Scale(SMA-FRS)
Change in Forced Vital Capacity | 22 months
  Forced Vital Capacity (FVC)
Change in Negative Inspiratory Force | 22 months
  Negative Inspiratory Force (NIF)
Change in lean muscle mass | 22 months
  Muscle mass measured using Dual-Energy X-Ray Absorptiometry (DXA)
Change in Quality of Life | 22 months
  Quality of life will be measured using 36-Item Short Form Survey (SF-36)
Change in Ulnar and Peroneal muscle measures | 22 months
  Compound Muscle Action Potential Amplitude (CMAP) will be recorded
Change in Motor Unit Number Estimation (MUNE) | 22 months
  Ulnar nerve (Recording at the Abductor Digiti Minimi muscle) MUNE scores will be recorded
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | 22 months
  Number of participants who experience adverse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Bakri Elsheikh, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States